CLINICAL TRIAL: NCT04320004
Title: Implementation and Evaluation of Clinic-based Medication Disposal Procedures to Reduce Unwanted and Unused Controlled Substances in Homes
Brief Title: Evaluation of a Medication Disposal Program in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Eric Wright, Professor, Geisinger Clinic
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-0606
Record Dates: First submitted 2020-03-18; First posted 2020-03-24 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Opioid-Related Disorders
Keywords: opioid; medication disposal; medication safety
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The investigators will use a cluster-randomized stepped-wedge design, using clinics as clusters (i.e., all clinics participate in all arms, but not all at the same time) to compare two main interventions (education only vs. education + mail-back bag) to baseline/usual care. In addition, the investigators will randomize patients in both intervention arms to receive or not to receive an added telephone reminder call through interactive voice response (IVR). The primary outcome of the study, medication disposal actions taken by the patient, will be assessed by a telephone survey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Baseline (No Intervention): Participating clinics will enter a baseline period where no interventions are used, but survey collection of baseline information about patient storage and disposal is collected. The baseline period varies depending on the cohort timing for each clinic but will last a minimum of one month for each clinic. In order to generate a survey list, the investigators will institute a "silent best practice alert (BPA)" in these clinics. This "Silent BPA" is not seen by providers, but a silent report is generated for reporting purposes, and for the study team to generate the baseline survey list.
- Education Intervention (Active Comparator): If a patient meets study criteria, an alert will fire in the EHR to remind the provider to discuss proper storage and disposal of the opioid medication with the subject. Following the subject's visit, participants will be mailed an education packet consisting of a cover letter and a flyer detailing the importance of medication disposal of unused opioids and instructing how to properly dispose. Between 30-45 days following the new opioid prescription, the survey call center will contact subjects by telephone to interview them regarding opioid prescription disposition and actions taken to disposal of any leftover medications, household information, their satisfaction with interventions, including provider-based education, and mailed educational material.
  Interventions: Behavioral: Education
- Education Intervention with Reminder (Active Comparator): This arm will follow the Education Intervention arm (BPA, provider education, mailed education and follow up survey) Approximately 50% of patients in the Education Intervention arm will be randomized to receive an interactive voice response (IVR) telephone call approximately 14 calendar days following receipt of his/her new opioid prescription. The IVR is intended to remind patients/caregivers to properly dispose of any unused medication and gather information from the patient on any disposal actions the patient has taken.
  Interventions: Behavioral: Education with Reminder
- Education + Disposal Bag Intervention (Active Comparator): If a patient meets study criteria, an alert will fire in the EHR to remind the provider to discuss proper storage and disposal of the opioid medication with the subject. Following the subject's visit, participants will be mailed an education packet consisting of a cover letter and a flyer detailing the importance of medication disposal of unused opioids and instructing how to properly dispose plus a postage paid medication disposal mail bag and instructions for use. Between 30-45 days following the new opioid prescription, the survey unit will contact subjects by telephone to interview them regarding opioid prescription disposition and actions taken to disposal of any leftover medications, household information, their satisfaction with interventions, including provider-based education, mailed educational material and mail-back bags.
  Interventions: Behavioral: Education + Disposal Bag
- Education + Disposal Bag Intervention with Reminder (Active Comparator): This arm will follow the Education+ Disposal Bag Intervention arm (BPA, provider education, mailed education+ disposal bag and follow up survey) Approximately 50% of patients in the Education + Disposal Bag Intervention arm will be randomized to receive an interactive voice response (IVR) telephone call approximately 14 calendar days following receipt of his/her new opioid prescription. The IVR is intended to remind patients/caregivers to properly dispose of any unused medication and gather information from the patient on any disposal actions the patient has taken.
  Interventions: Behavioral: Education + Disposal Bag with Reminder

INTERVENTIONS:
Behavioral: Education — Subject receives education
  Arms: Education Intervention
Behavioral: Education with Reminder — Subject receives education with reminder
  Arms: Education Intervention with Reminder
Behavioral: Education + Disposal Bag — Subject receives education and disposal bag
  Arms: Education + Disposal Bag Intervention
Behavioral: Education + Disposal Bag with Reminder — Subject receives education + disposal bag with reminder
  Arms: Education + Disposal Bag Intervention with Reminder

SUMMARY:
Evidence from recent trials primarily in the post-surgical patient population prescribed opioids for acute pain suggest patients more often properly dispose of unused opioids if instructed by a healthcare professional, if provided education on proper storage and disposal, and provided a physical medication disposal product (e.g. mail back bags). It is not clear how this evidence applied to patients in primary care will be readily adopted and sustained by practices and if the effectiveness will be comparable to that seen in other more controlled studies, largely limited to the surgical population. The objective of this trial is to evaluate a multifaceted program for safe medication disposal in primary care. Interventions include real-time best practice reminders to providers, educational materials mailed to patients, disposal mail-back bags supplied to patients and reminder phone calls. Proper medication disposal after 30 days following order will be assessed by telephone survey.

Our aims are to:

1. Evaluate a targeted intervention on patient's newly prescribed opioids within primary care.
2. Determine factors that influence patient action to remove unused opioid medications from the home.

DETAILED DESCRIPTION:
Prospective studies affirm that education and advice from providers to dispose of unused medications modestly improves medication disposal rates. Two recently published randomized controlled trials demonstrate improved disposal rates when a system for medication disposal, namely a medication disposal bag (e.g. return envelope or activated charcoal) were supplied to patients or caregivers. The impact of education and physical disposal mechanism inferred a greater magnitude of effect than education alone.

Research Design The investigators will use a cluster-randomized stepped-wedge design, using clinics as clusters (i.e., all clinics participate in all arms, but not all at the same time) to compare two main interventions (education only vs. education + mail-back bag). In addition, the investigators will randomize patients in both intervention arms to receive or not to receive an added telephone reminder call through interactive voice response (IVR). The primary outcome of the study, medication disposal actions taken by the patient, will be assessed by a telephone survey.

Study Population The investigators will enroll patients newly prescribed an opioid medication within one of the participating clinics. For patients younger than 18 years old, the investigators will follow clinic procedures for the engagement of parents or guardians; the investigators anticipate that management of medications in this population is largely handled by the guardian or parent and therefore these patients are of key interest when studying proper medication storage and disposal.

Interventions

(1) baseline; (2) education at the clinic level; (3) educational materials mailed to the patient's home; (4) mail back bags mailed to patient's homes and (5) IVR reminder calls

The study will enroll 13 clinics into the intervention with one clinic serving as an initial pilot. Feasibility and troubleshooting of the interventions will be tested within the pilot clinic; the pilot clinic will not be included within the final analysis.

All clinics will initially be assessed at baseline (usual care) followed by education only for approximately 3 months until the targeted quota of patients for the clinic is achieved. Following this attainment, new patients will begin receiving mail-back bags in addition to the education for the remainder of the enrollment period, in order to create the two main patient groups. Approximately 50% of patients during both education only and mail back bag stages of enrollment will be selected for IVR reminder calls, using a random number generator method.

Evaluation of safe medication disposal at 30-45 days post initial opioid prescription will be conducted through a telephone survey.

ELIGIBILITY:
Inclusion Criteria:

* Any patient receiving a new opioid prescription in a face-to-face or telehealth encounter in select Community Medicine Service Line practices.
* "New opioid prescription" is defined as a prescription for an opioid medication, Categories II-V (not anti-tussive) to a patient who has no opioid on current medication profile and no opioid prescriptions in the previous 3 months.
* Preferred language, as documented in the electronic health record (EHR), is English.
* Providers in participating primary care practices who receive the Best Practice Alert (BPA) for eligible patients.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1159 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Disposal of unused opioid following new opioid prescription | 30-45 days post new opioid prescription
  Proportion of patients with unused opioid medication who dispose opioid as assessed by telephone survey

SECONDARY OUTCOMES:
Patient satisfaction with medication mail back disposal bag | 30-45 days post new opioid prescription
  Patient satisfaction with mail-back bag, as assessed by telephone survey
Second prescription of opioid within 60 days post new opioid prescription | 60 days post new opioid prescription
  Prescription order for second opioid prescription as assessed by electronic health record

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wright, PharmD,MPH, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No